CLINICAL TRIAL: NCT00204620
Title: Multicenter Phase II Study With Bendamustin for Patients With Refractory Soft Tissue Sarcoma
Brief Title: Bendamustin Hydrochloride in Patients With Soft Tissue Sarcoma (STS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Arbeitsgemeinschaft fur Internistische Onkologie (Other); German Sarcoma Group (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: jth_002
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2007-04

CONDITIONS: Sarcoma, Soft Tissue
MeSH Terms: conditions — Sarcoma | interventions — Bendamustine Hydrochloride

INTERVENTIONS:
Drug: Bendamustin

SUMMARY:
The aims of this trial are to evaluate the efficacy of bendamustin in patients with metastatic soft tissue sarcoma who have progressed after or during an anthracycline-baesd chemotherapy and to assess the treatment of toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic or non-resectable soft tissue sarcoma
* Evidence of progression or relapse after an anthracycline-based and/ or ifosfamide-based chemotherapy
* At least 1 bidimensionally measurable tumor lesion according to RECIST criteria
* No previous radiation therapy on the only measurable lesion
* Willingness to receive regular follow-up
* Life expectancy more than 3 months
* ECOG status >= 2
* Patients aged 18 years and beyond
* leucocytes > 2500/µl, thrombocytes > 75000/µl)
* Serum creatine < 1,5 times the upper limit of normal value, GFR > 60/ml
* Written patient informed consent
* Ability to give informed consent

Exclusion Criteria:

* Previous or concurrent radiation of the index lesion (radiation of single lesion is allowed if not the index lesion)
* Insufficient liver function (bilirubin > 1.5 the upper limit of normal, prolongation of PT and aPTT > 1.5 the upper limit of normal; ASAT and ALAT > 3 the upper limit of normal (patients with liver metastases ASAT and ALAT > 5 the upper limit of normal)
* Active infection
* Prior therapy with Bendamustin hydrochloride
* Prior malignancies (other than adequately treated carcinoma in situ (CIS) of the cervix, bladder urothelium, basal cell carcinoma or adenoma of the colon including pTIS,pTIN), unless treated with curative intent and without evidence of disease > 5 years
* Symptomatic cardio- and/or cerebrovascular disease (NYHA-Scale III°)
* Interval since last chemotherapy < 4 weeks
* Evidence of CNS-metastases
* Evidence of pregnancy or lactation
* Woman of child-bearing potential without reliable methods of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28
Dates: Start 2002-03; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joerg T Hartmann, MD, Principal Investigator — South West German Cancer Center, Medical Center II, University of Tuebingen
Locations (1):
- Medical center II, University of Tuebingen, Tübingen, Germany